CLINICAL TRIAL: NCT00929630
Title: Seton or Glue for Trans-sphincteric Anal Fistulas. A Prospective Randomised Clinical Trial
Brief Title: Seton or Glue for Trans-sphincteric Anal Fistulas
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Evident advantages of one treatment (seton) over the other (Tissucol Glue)
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Donato F Altomare, Italian Society of Colorectal surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SICCR 10/2006
Record Dates: First submitted 2009-03-30; First posted 2009-06-29 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Anal Fistulas
Keywords: fibrin glue; transsphincteric anal fistulas; seton; incontinence; prospective randomised trial
MeSH Terms: conditions — Rectal Fistula | interventions — Adhesives; Fibrin Tissue Adhesive; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glue (Tissucol ) treatment (Experimental): patients with transsphincteric anal fistulas of cryptoglandular origin never operated on before
  Interventions: Procedure: glue (Tissucol) treatment; Procedure: Fistula closing with biological glue
- Seton treatment (Active Comparator): patients with transsphincteric anal fistulas of cryptoglandular origin never operated on before
  Interventions: Procedure: transsphincteric Seton positioning; Procedure: Seton positioning into the fistula tract

INTERVENTIONS:
Procedure: transsphincteric Seton positioning — A cutting seton is applied into the fistula tract
  Other Names: seton treatment of the fistula
  Arms: Seton treatment
Procedure: glue (Tissucol) treatment — After preparation of the fistula, a quantity of biological glue (Tissucol) is injected into the fistula tract
  Other Names: fibrin glue treatment of perianal fistulas
  Arms: glue (Tissucol ) treatment
Procedure: Fistula closing with biological glue — After cleaning and disinfection of the fistula tract, abot 1-2 ml of Tissucol (biological Glue) is inserted into the fistula tract to close it
  Other Names: fibrin glue treatment of perianal fistulas
  Arms: glue (Tissucol ) treatment
Procedure: Seton positioning into the fistula tract — Under spinal anesthesia a Seton is positioned into the fistula tract.
  Other Names: loose seton, cutting seton for anal fistulas
  Arms: Seton treatment

SUMMARY:
Surgical treatment of perianal fistulas frequently affects fecal continence. Sphincter saving techniques like loose or cutting seton and fistulectomy with advancement of an endorectal flap have been advocated to minimize the risk of sphincter injury, but patients often complain of a prolonged healing period and major discomfort. Furthermore, the healing rate varies widely according to the type of fistula and the surgeon's experience.In the early '90s the treatment of perianal fistulas by autologous or commercial fibrin glue was suggested and the American FDA approved the use and marketing of a human fibrin glue in 1998.

Since then, several studies have evaluated the effectiveness of human fibrin glue in the treatment of different types of perianal fistulas, reporting a wide range of success rates ranging from 31 to 85%.

Primary aim of this study is to conduct a prospective randomized trial evaluating the effectiveness of glue treatment of perianal fistulas as compared with the classical seton treatment. Secondary aims are to compare postoperative faecal incontinence, postoperative anal pain, healing time and length of hospitalization.

DETAILED DESCRIPTION:
Background: Fibrin glue treatment of anal fistulas has been proposed to minimize the risk of faecal incontinence but its acceptance by coloproctologists is still poor because clear data in literature are lacking. We will run a prospective randomised trial comparing commercial fibrin glue treatment with classical seton treatment, taking into account the healing rate, hospital stay, healing time, faecal incontinence and postoperative pain.

Patients and Methods: 130 homogeneous patients with trans-sphincteric anal fistulas referred to 7 Colorectal Units will be randomised to undergo fibrin glue or seton treatment. permanent healing of the fistula will be defined as absence on any discharge from the fistula and healing of the secondary fistula orifice after at least 1 year of follow up.

Post operative pain (on a VAS scale) and hospital stay will be recorded and compared in the two groups

ELIGIBILITY:
Inclusion Criteria:

* medium or high trans-sphincteric fistulas of cryptoglandular origin, no previous treatments

Exclusion Criteria:

* Crohn's disease
* anal abscesses
* complex fistulas (horse-shoe type or multiple secondary tracts)
* immunosuppression
* diabetes,
* anal fissures
* pregnancy
* anti-coagulant treatments,
* any allergic reaction to the bioglue components.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-01; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Fistula healing (absence of any discharge from the external fistula opening and complete healing of the external fistulas opening after at least 1 year of follow-up). The analysis of the population is not intention to treat. | 12 months

SECONDARY OUTCOMES:
Fecal continence and in-hospital stay | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Donato F Altomare, MD, Principal Investigator — University of Bari
Locations (1):
- Dept of Emergency and Organ transplantation - University of Bari, Bari, Italy